CLINICAL TRIAL: NCT03800680
Title: A Randomized Trial to Slow the Progression of Diabetes (The TRIPOD Study)
Brief Title: A Randomized Trial to Slow the Progression of Diabetes
Acronym: TRIPOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government); SingHealth Polyclinics (Other); Singapore General Hospital (Other); Changi General Hospital (Other)
Responsible Party: Principal Investigator, Eric A. Finkelstein, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HSRGDB16Dec003
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Smartphone application; Behavior change; Weight monitoring; Physical activity; Blood glucose monitoring; Medication adherence; Financial incentive; Cost-effectiveness analysis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Motor Activity; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (Arm 1) (No Intervention): Participants will receive usual care by their diabetes clinics.
- DMP (Arm 2) (Experimental): Participants will receive usual care by their diabetes clinics and the Diabetes Management Package (DMP).
  Interventions: Behavioral: Diabetes Management Package (DMP)
- DMP + M-POWER Rewards (Arm 3) (Experimental): Participants will receive usual care by their diabetes clinics, the Diabetes Management Package (DMP), and the financial incentive program, M-POWER Rewards.
  Interventions: Behavioral: Diabetes Management Package (DMP); Behavioral: M-POWER Rewards

INTERVENTIONS:
Behavioral: Diabetes Management Package (DMP) — M-POWER app: A one-stop portal to monitor diabetes self-management activities and progress. The app syncs and displays relevant data from study devices and apps.
  GlycoLeap: A 24-week, digitally-delivered education and behavior change program for T2DM patients.
  4 study devices with accompanying apps to aid in diabetes self-management: weighing scale, pedometer, glucometer, and pill tracker.
  Recommended activities:
  * Complete all 24 GlycoLeap lessons and quizzes
  * Weight Monitoring: Weigh at least once a week.
  * Physical Activity: At least 150 minutes of moderate-to-vigorous activity per week, targeting at least 420 Fitbit active minutes per week.
  * Blood Glucose Monitoring: At least three post-meal measurements within 4.0-10.0 mmol/L per week, with each reading taken on different days.
  * Medication: Take medications as prescribed.
  Arms: DMP (Arm 2); DMP + M-POWER Rewards (Arm 3)
Behavioral: M-POWER Rewards — A financial incentive program were participants can earn up to 516 M-Points (1 M-Point is equivalent to S$1) over the one-year study period for performing specific activities according to recommendations that are meant to improve glycemic control and for achieving HbA1c and weight loss goals. M-Points can be reimbursed in the form of financial rebates for approved non-inpatient healthcare-related expenses incurred during the study period.
  Arms: DMP + M-POWER Rewards (Arm 3)

SUMMARY:
The research objective of this one-year study is to test whether an evidence-based, low-cost mobile diabetes management package (DMP), with or without an incentive program grounded in economic theory (M-POWER Rewards), can effectively and cost-effectively improve health outcomes for adults with type 2 diabetes.

DETAILED DESCRIPTION:
Technological and economic advancement have created a major challenge to public health agencies in Singapore and other first world countries: the challenge being how to get individuals to maintain a healthy lifestyle when that is no longer a requirement for economic prosperity (and in fact may be a hindrance). What is required is a low cost strategy that effectively manages risk factors for chronic disease without overwhelming the public healthcare infrastructure. Although technology and economic advancement are clearly part of the problem, they may also be part of the solution.

For patients with type 2 diabetes mellitus (T2DM), lifestyle modification can be highly effective at stemming the progression of the disease. Effective interventions include modules that teach appropriate strategies for weight management, increased physical activity, better diet, routine glucose monitoring, and strict compliance to prescribed diabetes medications. These components can now be effectively delivered electronically. A recent review and meta-analysis of 13 smartphone applications for diabetes management found that these applications offered modest benefits, with a mean difference in HbA1c of -0.40%.

Because of the high costs involved in treating people with chronic conditions, employers, insurers, and governments all have a financial incentive to contain the chronic disease epidemic. Therefore, each has shown a willingness to invest in some level of prevention and treatment efforts. It is our contention that contingent rewards may be necessary to help people overcome their preferences for current over future consumption, often called present bias. Behavioral economists recommend that, to overcome present bias, rewards should be tied to both short-term and long-term outcomes or behaviors, such as monitoring blood glucose and taking medications as prescribed (short term) and pre-defined outcomes such as achieving a target HbA1c level over a specified duration (long term). Based on a recent systematic review of incentive studies conducted by members of our team, an optimal rewards strategy has the potential to greatly increase the effectiveness of existing mobile diabetes applications. If shown to be effective and cost effective, the investigators also believe payers will subsidize such a strategy.

Specifically, the investigators propose to conduct a 52-week, three-arm randomized controlled trial to evaluate whether an evidence-based, low-cost mobile diabetes management package (DMP), with or without an incentive program grounded in economic theory, can effectively and cost-effectively improve outcomes for adults with diabetes. The control arm (Arm 1) will receive usual care, whereas participants in the intervention arms will receive the DMP alone (Arm 2) or the DMP with the M-POWER Rewards incentive program (Arm 3) in addition to their usual care. The investigators hypothesize that participants in Arms 2 and 3 will show improved glycemic control, as measured by HbA1c levels, at the Month 12 primary endpoint compared to participants in the Arm 1 control group. The investigators also hypothesize that Arm 3 will have improved HbA1c levels compared to Arm 2 at Month 12. Similar hypotheses will be tested for secondary outcomes measured at Month 6.

In addition, the investigators will quantify the incremental cost-effectiveness of DMP with M-POWER Rewards and the net cost implications of both from a third party payer's perspective. The investigators hypothesize that despite its higher implementation cost, effectiveness will be greater and net cost will be lower for Arm 3 relative to the Arm 1 control group due to the reduction in medical expenditures that result from improved glycaemic control.

ELIGIBILITY:
All eligibility criteria will be self-declared.

Inclusion Criteria:

1. Diagnosed with T2DM with suboptimal diabetes control as defined by a HbA1c level of between 7.5% and 11.0% (inclusive) at their most recent test taken within the past six calendar months. This HbA1c inclusion criterion will be based on the patients' self-reported HbA1c levels and test dates.
2. Not on insulin.
3. On at least one oral glucose-lowering drug.
4. Singapore Citizen or Permanent Resident with no plans to relocate during the study period.
5. Able to read, write, and communicate in English.
6. Own a personal smartphone and be able to use it.

Exclusion Criteria:

1. Pregnant or lactating.
2. Diagnosed with chronic kidney disease (stage 3B with eGFR <45mL/min) or undergoing dialysis for end-stage kidney failure.
3. Diagnosed with liver cirrhosis.
4. Diagnosed with cancer that required treatment in the past five years.
5. Diagnosed with heart attack (i.e., acute myocardial infarction) within the past one year.
6. Diagnosed with heart failure (i.e., congestive heart failure)
7. Diagnosed with stroke or transient ischemic attacks.
8. Undergone whole blood or red blood cell transfusion within the past three months.
9. Diagnosed with severe anaemia (Haemoglobin <10g/dL)
10. Diagnosed with sickle-cell disease
11. Diagnosed with Thalassemia major
12. Undergone bariatric surgery or extensive bowel resection.
13. Undergone lower limb amputation (including toe amputation).
14. Taking systemic corticosteroids (including Traditional Chinese or Malay medicine).
15. Currently on doctor's advice against engaging in moderate-to-vigorous physical activity (i.e., brisk walking or more intense).
16. Currently have a condition(s) that restricts engaging in moderate-to-vigorous physical activity (i.e., brisk walking or more intense).

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2019-10-19 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-11 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c levels at Month 12 | Baseline, Month 12
  HbA1c or glycated hemoglobin is a measure of blood glucose levels. HbA1c blood tests will be conducted at baseline and Month 12 and the difference will be calculated.

SECONDARY OUTCOMES:
Change in HbA1c levels at Month 6 | Baseline, Month 6
  HbA1c or glycated hemoglobin is a measure of blood glucose levels. HbA1c blood tests will be conducted at baseline and Month 6 and the difference between the follow-up assessment (Months 6) and baseline will be calculated.
Change in weight at Months 6 and 12 | Baseline, Month 6, Month 12
  Weight will be measured at baseline, Month 6, and Month 12. The difference in weight between each follow-up assessment (Months 6 and 12) and baseline will be calculated.
Change in blood pressure at Months 6 and 12 | Baseline, Month 6, Month 12
  Blood pressure will be measured at baseline, Month 6, and Month 12. The difference in blood pressure between each follow-up assessment (Months 6 and 12) and baseline will be calculated.
Proportion of participants that had insulin treatment initiated by Months 6 and 12 | Baseline, Month 6, Month 12
  Percentage of participants that had insulin treatment initiated by their diabetes care physician by each follow-up assessment (Months 6 and 12).
Change in self-reported physical activity at Months 6 and 12 | Baseline, Month 6, Month 12
  Self-reported physical activity data will be collected at baseline, Month 6, and Month 12 via the Global Physical Activity Questionnaire (GPAQ). The difference in self-reported physical activity between each follow-up assessment (Months 6 and 12) and baseline will be calculated.
Change in self-reported weight monitoring at Months 6 and 12 | Baseline, Month 6, Month 12
  Self-reported weight monitoring data will be collected at baseline, Month 6, and Month 12. The difference in self-reported weight monitoring between each follow-up assessment (Months 6 and 12) and baseline will be calculated.
Change in self-reported blood glucose monitoring at Months 6 and 12 | Baseline, Month 6, Month 12
  Self-reported blood glucose monitoring data will be collected at baseline, Month 6, and Month 12. The difference in self-reported blood glucose monitoring between each follow-up assessment (Months 6 and 12) and baseline will be calculated.
Change in self-reported medication adherence at Months 6 and 12 | Baseline, Month 6, Month 12
  Self-reported medication adherence data will be collected at baseline, Month 6, and Month 12. The difference in self-reported medication adherence between each follow-up assessment (Months 6 and 12) and baseline will be calculated.
Change in self-reported diabetes self-management at Months 6 and 12 | Baseline, Month 6, Month 12
  Self-reported diabetes self-management data will be collected at baseline, Month 6, and Month 12 via the Diabetes Self-Management Questionnaire (DSMQ). The difference in self-reported diabetes self-management between each follow-up assessment (Months 6 and 12) and baseline will be calculated.
Change in self-reported sleep quality at Months 6 and 12 | Baseline, Month 6, Month 12
  Self-reported sleep quality data will be collected at baseline, Month 6, and Month 12 via the Pittsburgh Sleep Quality Index (PSQI). The difference in self-reported sleep quality between each follow-up assessment (Months 6 and 12) and baseline will be calculated.
Change in self-reported work productivity and daily activity impairment at Months 6 and 12 | Baseline, Month 6, Month 12
  Self-reported work productivity and daily activity impairment data will be collected at baseline, Month 6, and Month 12 via a modified Work Productivity and Activity Impairment: Specific Health Problem instrument (WPAI:SHP). The difference in self-reported work productivity and daily activity impairment between each follow-up assessment (Months 6 and 12) and baseline will be calculated.
Change in self-reported health utility index at Months 6 and 12 | Baseline, Month 6, Month 12
  Self-reported health utility index data will be collected at baseline, Month 6, and Month 12 via the EQ-5D-5L questionnaire. The difference in self-reported health utility index between each follow-up assessment (Months 6 and 12) and baseline will be calculated.
Incremental cost-effectiveness ratios based on HbA1c at Month 12 | Baseline, Month 12
  Incremental cost-effectiveness ratios will be determined by calculating the incremental cost per unit reduction in HbA1c at Month 12 (primary endpoint) compared to baseline.
Incremental cost-effectiveness ratios based on QALY at Month 12 | Baseline, Month 12
  Incremental cost-effectiveness ratios will be determined by calculating the incremental cost per quality adjusted life year (QALY) gained at Month 12 (primary endpoint) compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Finkelstein, PhD, MHA, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Duke-NUS Medical School, Singapore, Singapore

REFERENCES:
- [Derived] Bairavi J, Gardner DS, Yeoh E, Tham KW, Gandhi M, Tan NC, Lee PC, Lim RSM, Adamjee T, Cheung YB, Bee YM, Finkelstein EA. Protocol update and baseline characteristics for the TRIal to slow the Progression of Diabetes (TRIPOD) randomized controlled trial. Trials. 2023 Nov 14;24(1):728. doi: 10.1186/s13063-023-07770-7. PMID 37964330
- [Derived] Lim RSM, Gardner DSL, Bee YM, Cheung YB, Bairavi J, Gandhi M, Goh SY, Ho ETL, Lin X, Tan NC, Tay TL, Finkelstein EA. TRIal to slow the Progression Of Diabetes (TRIPOD): study protocol for a randomized controlled trial using wireless technology and incentives. Trials. 2019 Nov 28;20(1):650. doi: 10.1186/s13063-019-3749-x. PMID 31779678